CLINICAL TRIAL: NCT01916564
Title: Efficacy and Tolerability of Split-dose Versus Same-day Administration of Reduced-volume PEG-ELS Plus Bisacodyl for Morning Colonoscopy: a Randomised Trial
Brief Title: Split-dose Versus Same-day Reduced-volume PEG-ELS Plus Bisacodyl for Morning Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Chan Wah Kheong, Senior Lecturer and Consultant Gastroneterologist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SplitAMBPrep
Record Dates: First submitted 2013-07-26; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Bowel Preparation for Morning Colonoscopy
Keywords: Bowel preparation; Morning colonoscopy; Split-dose; Same-morning whole-dose; Reduced-volume PEG-ELS

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Same-morning whole-dose (Active Comparator): 2-L PEG-ELS between 5 a.m. and 6 a.m. on the day of colonoscopy
  Interventions: Other: Same-morning whole-dose
- Split-dose (Active Comparator): 1-L PEG-ELS between 8 p.m. and 8.30 p.m. on the day before and 1-L PEG-ELS between 5.30 a.m. and 6 a.m. on the day of colonoscopy
  Interventions: Other: Split-dose

INTERVENTIONS:
Other: Split-dose — 2 tablets of bisacodyl 5 mg at 8 p.m. two days before colonoscopy
  Low fibre diet and 2 tablets of bisacodyl 5 mg at 8 p.m. on the day before colonoscopy
  1-L PEG-ELS between 8 p.m. and 8.30 p.m. on the day before and 1-L PEG-ELS between 5.30 a.m. and 6 a.m. on the day of colonoscopy
  Arms: Split-dose
Other: Same-morning whole-dose — 2 tablets of bisacodyl 5 mg at 8 p.m. two days before colonoscopy
  Low fibre diet and 2 tablets of bisacodyl 5 mg at 8 p.m. on the day before colonoscopy
  2-L PEG-ELS between 5 a.m. and 6 a.m. on the day of colonoscopy
  Arms: Same-morning whole-dose

SUMMARY:
This study aims to compare split-dose vs. same-morning whole-dose of 2-litre PEG-ELS plus bisacodyl for bowel preparation for morning outpatient colonoscopy.

DETAILED DESCRIPTION:
A good bowel preparation regime is one that is not only effective in cleansing the colon but should be relatively small in volume and well-tolerated by patients with minimal adverse gastrointestinal symptoms. At our centre, reduced-volume 2-litre PEG-ELS plus bisacodyl and low fiber diet is used for bowel preparation for patients undergoing colonoscopy. Patients undergoing morning outpatient colonoscopy would normally ingest the PEG-ELS and bisacodyl the day before. This regime has been shown to be better tolerated by patients without compromising the quality of bowel preparation when compared with conventional 4-liter PEG-ELS. However, previous study on patient satisfaction found that nearly half of the patients attending the outpatient colonoscopy service at our centre were dissatisfied with the bowel preparation regime used. Of the seven items considered in the evaluation of patient satisfaction, comfort level during bowel preparation was the main cause of unfavorable responses. Moreover, a separate study using the same bowel preparation regime at our centre found a high percentage of poor quality bowel preparation, which was associated with increased technical difficulty and patient discomfort during colonoscopy. There was clearly a need for a better bowel preparation regime. Current literature suggests that either taking reduced-volume PEG-ELS on the same morning instead of the previous evening, or splitting the bowel preparation, would be better. However, whether the former or the latter is better, is unknown. The aim of our study was to compare the use of same-morning whole-dose reduced-volume PEG-ELS and split-dose reduced-volume PEG-ELS for bowel preparation for patients undergoing morning outpatient colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients undergoing morning outpatient colonoscopy at the Endoscopy Unit, University of Malaya Medical Centre

Exclusion Criteria:

* In-patients, patients scheduled for afternoon colonoscopy, patients who used other bowel preparation regime than that assigned, patients who had incomplete examination not related o quality of bowel preparation e.g. obstructing tumour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | During the colonoscopy procedure itself which spans an average of 20 minutes
  Using the Boston Bowel Preparation Scale and an overall grading by the endoscopist
Patient tolerability | The period from commencement of bowel preparation to the colonoscopy procedure itself which spans approximately 36 hours
  Using the questionnaire by Aronchick and colleagues and an ordinal five-value Likert scale question on comfort level during bowel preparation

SECONDARY OUTCOMES:
Technical aspects of colonoscopy | During the colonoscopy procedure itself which spans an average of 20 minutes
  Cecal intubation rate, cecal intubation, withdrawal and colonoscopy times, adenoma detection rate and number of adenoma detected are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Wah Kheong Chan, Principal Investigator — University of Malaya
Locations (1):
- Endoscocpy Unit, University of Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Chan WK, Azmi N, Mahadeva S, Goh KL. Split-dose vs same-day reduced-volume polyethylene glycol electrolyte lavage solution for morning colonoscopy. World J Gastroenterol. 2014 Oct 21;20(39):14488-94. doi: 10.3748/wjg.v20.i39.14488. PMID 25339836